CLINICAL TRIAL: NCT01727661
Title: Cardiopulmonary Fitness, Lung Function, Muscular Oxygen Saturation, and Quality of Life in Patients With Type 1 Diabetes Mellitus
Brief Title: Cardiopulmonary Fitness, Lung Function, Muscular Oxygen Saturation, and Quality of Life in T1DM
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201201005RIC
Record Dates: First submitted 2012-07-08; First posted 2012-11-16 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: diabetes mellitus; cardiopulmonary fitness; lung function; muscular oxygenation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Exercise Test; Spectroscopy, Near-Infrared; Quality of Life

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- type 1 diabetes mellitus: 1. exercise testing with near-infrared spectroscopy
  2. lung function testing
  3. quality of life
  Interventions: Behavioral: exercise testing with near-infrared spectroscopy; Behavioral: lung function testing; Behavioral: quality of life
- healthy controls: 1. exercise testing with near-infrared spectroscopy
  2. lung function testing
  3. quality of life
  Interventions: Behavioral: exercise testing with near-infrared spectroscopy; Behavioral: lung function testing; Behavioral: quality of life

INTERVENTIONS:
Behavioral: exercise testing with near-infrared spectroscopy — subjects will sit on the ergometer, resting heart rate and BP will be measured for at least 2 minutes. Before testing, each participant will be informed to perform cycling with 0 watt for 2 minutes. Then, exercise testing will be started at 30 watt, and increase 15 watt in male and 10 watt in female every minute until the termination criteria achieved.
Behavioral: lung function testing — spirometry testing: Each participant will then place mouthpiece in mouth and close lips around the mouthpiece. Participants will inhale completely and rapidly and then exhale maximally until no more air could be expelled while maintaining an upright position. Values of FEV1 (forced expiratory volume in 1 second) and FVC (forced vital capacity) will be calculated immediately after the exhalation.
  single-breath carbon monoxide diffusing capacity: Participants will sit on a firm and nose clips will then be attached and mouthpiece be placed in mouth. After participants perform several stable breathes, testing starts with a complete exhalation. Each participant will be instructed to inhale rapidly and completely and then hold for 10 seconds.
Behavioral: quality of life — assessing quality of life using short-forum 36 (questionnaire)

SUMMARY:
The purpose of this study is to compare the differences of

1. cardiopulmonary fitness
2. lung function
3. muscular oxygen saturation
4. quality of life between type 1 diabetes mellitus and healthy adults.

DETAILED DESCRIPTION:
This study is also to investigate the relationships between cardiopulmonary fitness, lung function, muscular oxygen saturation, glycemic control, and quality of life in patients with type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 1 diabetes mellitus ≥2 years (diabetic group)
* age-, gender-, and BMI-matched healthy subjects (control group)

Exclusion Criteria:

* cardiac or respiratory disease
* pregnancy
* hospitalization due to any medical condition in recent 6 months
* any other condition affecting exercise performance or lung function.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: outpatient department
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
exercise testing with near-infrared spectroscopy | at baseline

SECONDARY OUTCOMES:
lung function | at baseline
  flow volume loop, lung diffusing capacity
quality of life | at baseline
  short-forum 36

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Tai Wu, phD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Wanke T, Formanek D, Auinger M, Zwick H, Irsigler K. Pulmonary gas exchange and oxygen uptake during exercise in patients with type 1 diabetes mellitus. Diabet Med. 1992 Apr;9(3):252-7. doi: 10.1111/j.1464-5491.1992.tb01771.x. PMID 1576807
- [Background] Komatsu WR, Barros Neto TL, Chacra AR, Dib SA. Aerobic exercise capacity and pulmonary function in athletes with and without type 1 diabetes. Diabetes Care. 2010 Dec;33(12):2555-7. doi: 10.2337/dc10-0769. Epub 2010 Aug 31. PMID 20807874